CLINICAL TRIAL: NCT03087630
Title: Informing Alcohol-Related Risk Intervention With the Prototype Willingness Model: Evaluating Personalized Information and Choices
Brief Title: Evaluating Personalized Information and Choices
Acronym: EPIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Melissa Lewis, Professor, Psychiatry and Behavioral Sciences, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 44051
Record Dates: First submitted 2017-03-08; First posted 2017-03-22 (Actual); Last update posted 2018-05-18 (Actual); Status verified 2018-05

CONDITIONS: Feedback, Psychological; Underage Alcohol Use; Risk-Taking; Sex Behavior
MeSH Terms: conditions — Underage Drinking; Risk-Taking; Sexual Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Reasoned-Based Intervention (Experimental): Receives reason-based intervention.
  Interventions: Behavioral: Reasoned-Based Intervention
- Social-Based Intervention (Experimental): Receives social-based intervention.
  Interventions: Behavioral: Social-Based Intervention
- Integrated Intervention (Experimental): Receives integrated intervention.
  Interventions: Behavioral: Integrated Intervention
- Attention Control (Experimental): Receives attention control feedback.
  Interventions: Behavioral: Attention Control

INTERVENTIONS:
Behavioral: Reasoned-Based Intervention — Receives personalized feedback based on the reasoned pathway of the Prototype Willingness Model.
  Arms: Reasoned-Based Intervention
Behavioral: Social-Based Intervention — Receives personalized feedback based on the social pathway of the Prototype Willingness Model.
  Arms: Social-Based Intervention
Behavioral: Integrated Intervention — Receives personalized feedback based on both the reasoned and social pathways of the Prototype Willingness Model.
  Arms: Integrated Intervention
Behavioral: Attention Control — Receives personalized feedback related to nutrition and exercise, unrelated to drinking behavior.
  Arms: Attention Control

SUMMARY:
This research examines a theoretically informed web-based personalized feedback intervention to reduce alcohol-related risky sexual behavior among young adult drinkers. To accomplish this objective the study has enrolled a national sample of 1200 young adults aged 18-20 and is in the process of assessing them at 3-, 6-, 9-, and 12-months. The investigators will evaluate the overall efficacy of the interventions based on the Prototype Willingness Model by comparing underage young adult drinkers randomly assigned to receive the reason-based pathway intervention (n=300), the social-based pathway intervention (n=300), or the integrated intervention based on the full Prototype Willingness Model (both pathways, n=300) to an attention control group (n=300). The investigators will examine whether changes in components of both the reasoned and social pathways and drinking mediate intervention efficacy on reducing alcohol-related risky sexual behavior. Past behavior and college student status will be evaluated as moderators of intervention efficacy. The proposed study is both significant and innovative in that it will evaluate brief interventions among a national sample of young adults attending and not attending college, will utilize social networking sites for participant recruitment, and will test the efficacy of interventions based on individual and integrated pathways of the Prototype Willingness Model.

DETAILED DESCRIPTION:
Purpose

This research is designed to evaluate a personalized feedback intervention for alcohol-related risky sexual behavior in a longitudinal study of underage young adult drinkers aged 18-20. The intervention is theoretically based on the Prototype Willingness Model (PW Model). The Prototype Willingness Model assumes two pathways to risk behavior: one pathway that is reasoned and one pathway that is socially based. Prior research has shown that interventions consistent with, or based on, components of the Prototype Willingness Model, are efficacious at reducing alcohol use and risky sexual behavior.

The investigators will evaluate the overall efficacy of the interventions based on the PW Model by comparing underage young adult drinkers randomly assigned to receive the reasoned-based pathway intervention (n=300), the social-based pathway intervention (n=300), or the integrated intervention based on the full PW Model (both pathways; n=300) to an attention control group (n=300). The investigators will examine whether intervention efficacy at reducing alcohol-related risky sexual behavior is mediated by reductions in drinking and changes in components of both the reasoned and social pathways (e.g., changes in attitudes, injunctive and descriptive normative perceptions, behavioral intention, perceived vulnerability, prototype favorability, and behavioral willingness). Past behavior and college student status will be evaluated as moderators of intervention efficacy. The investigators will also examine whether effects of all three interventions are maintained across the study follow-up period.

Procedures

This study consists of two phases. Phase 1 consists of a one-time online survey for the purpose of collecting normative data to be used in the personalized feedback intervention in Phase 2. Phase 2 will include an online screening, baseline assessment, and personalized feedback intervention, followed by four follow-up assessments.

Initial recruitment procedures for Phase 1 and 2 follow the same protocol. In both phases, young people who view study advertisements and choose to log-on to the study website view a brief information statement and, upon providing consent, proceed to a brief online screening survey containing questions regarding their basic demographics and contact information and questions necessary for determining eligibility, detailed below. Those who complete the survey and meet online eligibility are told that participants will be contacted by phone within 3 business days by research staff to explain the study and determine eligibility (e.g., age verification). During the 5 minute telephone screen, potential participants are given more information about the study and have their age verified by research staff. Previously reported demographics (age, DOB, etc.) from the online screening survey are cross checked for data consistency. Once investigators verify age and other screening criteria participants are given the option to receive a link via e-mail with more information about the study (i.e., information statement) and to participate in the web-survey. Upon completion of the telephone screen, interested and eligible participants are emailed a link to the one-time assessment (for Phase 1) or the baseline assessment (for Phase 2), as well as a unique PIN in a separate email. Each of these surveys begins with a full information statement, to which participants can indicate consent and begin the assessment. Those who begin but do not complete the assessment are contacted via email and telephone. If at any time a participant indicates unwillingness to continue, no further contact will ensue.

The Phase 1 one-time assessment is a 30-45-minute survey which consists of questions focusing on alcohol-related risky sexual behavior and injunctive and descriptive normative perceptions regarding alcohol-related risky sex behavior in others. Participants who complete this assessment are paid with a gift certificate, emailed within 2 weeks of completing the survey.

For Phase 2, the 30-45-minute baseline survey will consist of questions similar to the Phase 1 survey. Upon completion of the baseline assessment, participants will be randomized to one of four conditions: reasoned-based pathway intervention (n=300), social-based pathway intervention (n=300), integrated intervention (based on both pathways; n=300), or an attention control group (n=300). Participants randomized to an intervention condition will receive web-based graphic personalized feedback that will be imbedded into an interactive web-based assessment. The control condition will receive attention control feedback. The feedback is non-confrontational in tone, seeks to increase motivation to reduce alcohol-related risky sexual behavior, and is based on information provided during the baseline assessment. Participants will be able to view the feedback online and print it after viewing the entire feedback, or can click to request that a copy be mailed to them. All personalized feedback interventions will be tailored based on sexual orientation where appropriate.

Follow-up assessments will occur 3, 6, 9, and 12 months after baseline and will follow the same protocol and include the same measures. Participants will be emailed an invitation with a link to the survey and a separate PIN email

Participants will be paid with gift certificate for each assessment completed, and will also be eligible for entry into a drawing at each assessment. Gift certificates will be e-mailed to the participant within 2 weeks of completing the survey.

Subjects

Phase 1 Participants will include approximately 1,000 young adults aged 18-20, who live in the United States and who complete a one-time online assessment.

Phase 2 Participants will include 1,200 young adults aged 18-20, who live in the United States and who complete the baseline survey.

ELIGIBILITY:
Study 1 Inclusion & Exclusion Criteria

Inclusion Criteria:

* 18-20 years old
* Not in high school
* Reside within the US
* Have a valid email address

Exclusion Criteria:

* There are no exclusion criteria other than not meeting inclusion criteria

Study 2 Inclusion & Exclusion Criteria

Inclusion Criteria:

* 18-20 years old
* Not in high school
* Reside within the US
* Have a valid email address
* Not currently in monogamous relationship
* Drink at least two times per week
* Have had sex at least once within the past 3 months
* Did not participate in Phase 1

Exclusion Criteria:

* There are no exclusion criteria other than not meeting inclusion criteria

Ages: 18 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1204 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2018-03-26 (Actual); Study Completion 2018-03-26 (Actual)

PRIMARY OUTCOMES:
Change in Frequency of Drinking Prior to Sex | Baseline, 3-, 6-, 9-, and 12-Month Follow-Ups
  Assesses frequency of drinking prior to sex at the baseline, 3-, 6-, 9-, and 12-month time points.
Change in Typical Number of Drinks Consumed Prior to Sex | Baseline, 3-, 6-, 9-, and 12-Month Follow-Ups
  Assesses typical number of drinks consumed prior to sex at the baseline, 3-, 6-, 9-, and 12-month time points.
Change in Total Number of Sex Partners Involving Alcohol | Baseline, 3-, 6-, 9-, and 12-Month Follow-Ups
  Assesses total number of sex partners involving alcohol at the baseline, 3-, 6-, 9-, and 12-month time points.
Change in Total Number of Casual Sex Partners Involving Alcohol | Baseline, 3-, 6-, 9-, and 12-Month Follow-Ups
  Assesses total number of casual sex partners involving alcohol at the baseline, 3-, 6-, 9-, and 12-month time points.
Change in Frequency of Condom Use During Sex Involving Alcohol | Baseline, 3-, 6-, 9-, and 12-Month Follow-Ups
  Assesses frequency of condom use during sex involving alcohol at the baseline, 3-, 6-, 9-, and 12-month time points.

IPD SHARING:
Plan to Share IPD: No
A select number of researchers will have access to unidentified participant data at the close of the study.